CLINICAL TRIAL: NCT03724162
Title: Impact of Circulatory Changes on Thoracic Anastomosis in Patients Undergoing Thoracolaparoscopic Surgery for Oesophageal Carcinoma
Brief Title: Evaluation of the Circulatory Status of Stomach Tube and Gastrooesophageal Anastomosis
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Syed Sajid Hussain Kazmi, Consultat Vascular Surgeon, Oslo University Hospital
Other Study IDs: LDFLVS Ca oesophagus
Record Dates: First submitted 2018-07-26; First posted 2018-10-30 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Circulatory; Change; Microcirculation
Keywords: cancer oesophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of anastomotic leaks after gastroesophageal anastomosis after thoracolaparoscopic cancer esophagus surgery is high at the Oslo University Hospital. The patients selected for operation shall be investigated for microcirculatory changes at the thoracic anastomosis site and followed up for any post operative anastomotic leaks.

DETAILED DESCRIPTION:
- Microcirculation shall be evaluated during the operation with trans serosal laser doppler flowmetry and visible light spectroscopy (LDFVLS). Different anatomical areas of the stomach and gastric tube shall be examined With LDFVLS to find any changes in SO2, rHb, flow, and velocity. Repeat measurements shall be taken to compare them with the baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

Patients with oesophageal carcinoma planned to have thoracolaparoscopic operation and thoracic gastroesophageal anastomosis shall be included.

Exclusion Criteria: Patients who do not give written consent will not be included.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Only subjects selected for thoracolaparoscopic operation shall be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Impact of local microcirculatory changes on the thoracooesophegial anastomosis after cancer oesophagus surgery | 6 months
  Repeated measurements of microcirculation With laser dopper flometer and visible light spectrometry shall be performed trans serosally of the stoach and gastric tube to register changes in microcirculation. Patients shall be followed up for anastomotic leaks. Besides CT angiography shall be performed before surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo
  - Department of vascular surgery, Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No